CLINICAL TRIAL: NCT02475135
Title: A Single-dose, Open-label, Randomized, Crossover Study to Assess the Impact of Food on the Pharmacokinetics of Darunavir, Cobicistat, Emtricitabine, and Tenofovir Alafenamide Administered as a Fixed-dose Combination Tablet, and the Relative Bioavailability
Brief Title: Relative Bioavailability and Food Effect for Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Fixed Dose Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR107430; 2015-001213-27 (EudraCT Number); TMC114FD2HTX1002 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2015-06-15; First posted 2015-06-18 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Immunodeficiency Virus Type 1, Human; Immunodeficiency Virus Type 2, Human; Darunavir; Cobicistat; Tenofovir Alafenamide; Emtricitabine; Elvitegravir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; elvitegravir; Cobicistat; Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Panel 1: Group 1 (Experimental): Subject will receive a single oral tablet of fixed dose combination (FDC) containing darunavir (DRV)/ cobicistat (COBI)/emtricitabine (FTC) /tenofovir alafenamide (TAF) (D/C/F/TAF) under fed conditions (standardized regular breakfast, test Panel 1) on Day 1 of treatment period 1 and by FDC of elvitegravir (EVG)/cobicistat (COBI)/emtricitabine (FTC)/ tenofovir alafenamide (TAF) (E/C/F/TAF) under fed conditions (standardized regular breakfast, reference Panel 1) on Day 1 of treatment period 2.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Drug: Elvitegravir /Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Other: Standardized Regular Breakfast
- Panel 1: Group 2 (Experimental): Subject will receive a single oral tablet of FDC containing E/C/F/TAF under fed conditions (standardized regular breakfast, reference Panel 1) on Day 1 of treatment period 1 and a single oral tablet of FDC containing D/C/F/TAF under fed conditions (standardized regular breakfast, test Panel 1) on Day 1 of treatment period 2.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Drug: Elvitegravir /Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Other: Standardized Regular Breakfast
- Panel 2: Group 1 (Experimental): Subject will receive a single oral tablet of D/C/F/TAF under fed conditions (standardized regular breakfast, test Panel 2) on Day 1 of treatment period 1 and a single oral tablet of DRV, a tablet of emtricitabine/ tenofovir alafenamide (FTC/TAF) and a tablet of COBI under fed conditions (standardized regular breakfast, reference Panel 2) on Day 1 of treatment period 2.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Drug: Darunavir; Drug: Emtricitabine/Tenofovir alafenamide (FTC/TAF); Drug: Cobicistat; Other: Standardized Regular Breakfast
- Panel 2: Group 2 (Experimental): Subject will receive a single oral tablet of DRV, a tablet of FTC/TAF and a tablet of COBI under fed conditions (standardized regular breakfast, reference Panel 2) on Day 1 of treatment period 2 and a single oral tablet of D/C/F/TAF under fed conditions (standardized regular breakfast, test Panel 2) on Day 1 of treatment period 2.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Drug: Darunavir; Drug: Emtricitabine/Tenofovir alafenamide (FTC/TAF); Drug: Cobicistat; Other: Standardized Regular Breakfast
- Panel 3: Group 1 (Experimental): Subject will receive a single oral tablet of D/C/F/TAF under fasted conditions (test Panel 3) on Day 1 of treatment period 1 and a single oral tablet of D/C/F/TAF with a standardized high-fat breakfast (reference Panel 3) on Day 1 of treatment period 2.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC
- Panel 3: Group 2 (Experimental): Subject will receive a single oral tablet of D/C/F/TAF with a standardized high-fat breakfast (reference Panel 3) on Day 1 of treatment period 1 followed by a single oral tablet of D/C/F/TAF under fasted conditions (test Panel 3) on Day 1 of treatment period 2.
  Interventions: Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC; Other: High-fat Breakfast

INTERVENTIONS:
Drug: Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide FDC — A tablet containing DRV 800 mg, COBI 150 mg, FTC 200 mg and TAF 10 mg as FDC will be administered.
Drug: Elvitegravir /Cobicistat/Emtricitabine/Tenofovir alafenamide FDC — A tablet containing EVG 150 mg, COBI 150 mg, FTC 200 mg and TAF 10 mg as FDC will be administered.
  Arms: Panel 1: Group 1; Panel 1: Group 2
Drug: Darunavir — A tablet containing Darunavir (DRV) 800 mg will be administered.
  Arms: Panel 2: Group 1; Panel 2: Group 2
Drug: Emtricitabine/Tenofovir alafenamide (FTC/TAF) — A tablet containing Emtricitabine (FTC) 200 mg and Tenofovir alafenamide (TAF) 10 mg will be administered.
  Arms: Panel 2: Group 1; Panel 2: Group 2
Drug: Cobicistat — A tablet containing cobicistat (COBI) 150 mg will be administered.
  Arms: Panel 2: Group 1; Panel 2: Group 2
Other: High-fat Breakfast — High-fat breakfast will be administered.
  Arms: Panel 3: Group 2
Other: Standardized Regular Breakfast — Standardized regular breakfast will administered.
  Arms: Panel 1: Group 1; Panel 1: Group 2; Panel 2: Group 1; Panel 2: Group 2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and relative bioavailability of Emtricitabine (FTC) and Tenofovir alafenamide (TAF) when administered as a fixed-dose combination (FDC) with darunavir (DRV) and cobicistat (COBI) (darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) relative to administration as an FDC with Elvitegravir (EVG) and COBI (Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide), under fed conditions in healthy subjects (Panel 1); evaluate the single-dose pharmacokinetics and relative bioavailability of DRV, COBI, FTC and TAF when administered as an FDC (D/C/F/TAF) or as separate agents (D+C+FTC/TAF), under fed conditions in healthy subjects (Panel 2) and to evaluate the impact of food (fasting or high-fat breakfast) on the single-dose pharmacokinetics of DRV, COBI, FTC, and TAF when administered as an FDC (D/C/F/TAF) in healthy subjects (Panel 3).

DETAILED DESCRIPTION:
This is a Phase 1, 3-panel, open-label, randomized, 2-way crossover study in healthy subjects. Healthy subjects will be divided over 3 panels (Panel 1, 2 and 3). Subjects will be randomized within each panel. In each panel, during 2 subsequent sessions, each subject will receive 2 treatments (Treatments A and B in Panel 1, Treatments C and D in Panel 2, and Treatments E and F in Panel 3). Each treatment is defined as follows: Treatment A: single oral dose of D/C/F/TAF 800/150/200/10 milligram (mg) as FDC tablet under fed conditions (standardized regular breakfast); Treatment B: single oral dose of E/C/F/TAF 150/150/200/10 mg as FDC tablet under fed conditions; Treatment C: single oral dose of D/C/F/TAF 800/150/200/10 mg as FDC tablet under fed conditions; Treatment D: single oral dose of DRV as 800-mg tablet, FTC/TAF as 200/10 mg tablet and COBI 150 mg tablet under fed conditions. Treatment E: single oral dose of D/C/F/TAF 800/150/200/10 mg as FDC tablet, under fasted condition and Treatment F: single oral dose of D/C/F/TAF 800/150/200/10 mg tablet, with a standardized high-fat breakfast. Each treatment will be separated by a washout period of at least 7 days. Primarily pharmacokinetic parameters will be assessed. Subjects' safety will be assessed throughout.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a non-smoker for at least 3 months prior to selection
* Subject must have a body mass index (BMI, weight in kg divided by the square of height in meters) of 18.5 to 30.0 kg/m^2, extremes included
* Subject must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead ECG performed at screening. If the results are outside the normal reference ranges, the subject may be included only if they are not listed under the exclusion criteria and if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the subject's source documents and initialed by the Investigator
* Subject must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the biochemistry panel, hematology, or urinalysis are outside the normal reference ranges, the subject may be included only if the abnormalities or deviations from normal are not listed in the exclusion criteria, and the Investigator judges they are not clinically significant. This determination must be recorded in the subject's source documents and initialed by the Investigator
* Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Subject has a positive human immunodeficiency virus-1 (HIV-1) or HIV-2 test at screening
* Subject has hepatitis A, B, or C infection (confirmed by a positive hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen, and/or hepatitis C virus antibody, respectively) at screening
* Subject has currently significant and active diarrhea, nausea, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability
* Subject has any history of renal insufficiency
* Subject has known allergies, hypersensitivity, or intolerance to DRV, COBI (GS-9350), EVG (Panel 1 only), FTC, TAF or their excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-08-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events | From signing the Informed Consent Form (ICF) up to 10 days after last study drug administration
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

OTHER OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Plasma Concentration at the Last Quantifiable Time Point (Clast) of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The Clast is the last observed quantifiable plasma concentration above the quantification limit.
Elimination Rate Constant (Lambda[z]) of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time to Last Quantifiable Plasma Concentration (Tlast) of Darunavir (DRV), cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  The Tlast is the time to last observed quantifiable plasma concentration.
Ratio of AUClast of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  Ratio of individual AUClast values between test and reference treatment will be observed. For Panel 1, test will be treatment A and reference will be treatment B, for Panel 2, test will be treatment C and reference will be treatment D and for Panel 3, test will be treatment D and reference will be treatment F.
Ratio of AUC[0-infinity] of Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC) and Tenofovir Alafenamide (TAF) | Up to 72 Hours after study drug administration
  Ratio of individual AUC[0-infinity] values between test and reference treatment will be observed. For Panel 1, test will be treatment A and reference will be treatment B, for Panel 2, test will be treatment C and reference will be treatment D and for Panel 3, test will be treatment D and reference will be treatment F.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trials, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Antwerp, Belgium

REFERENCES:
- [Derived] Crauwels HM, Baugh B, Van Landuyt E, Vanveggel S, Hijzen A, Opsomer M. Bioequivalence of the Once-Daily Single-Tablet Regimen of Darunavir, Cobicistat, Emtricitabine, and Tenofovir Alafenamide Compared to Combined Intake of the Separate Agents and the Effect of Food on Bioavailability. Clin Pharmacol Drug Dev. 2019 May;8(4):480-491. doi: 10.1002/cpdd.628. Epub 2018 Nov 9. PMID 30412360